CLINICAL TRIAL: NCT01770158
Title: Maintenance Therapy With Histamine Dihydrochloride and Interleukin-2 in Adult Acute Myeloid Leukemia (AML) Patients With Measurable Minimal Residual Disease (MRD)- a Non-interventional Study (NIS)
Status: Terminated | Type: Observational
Why Stopped: Recruitment goal cannot be achieved any more as only 8 patients have been recruited since start of the study in 2012.
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Jochen Greiner, Prof. Dr. Jochen Greiner, University of Ulm
Other Study IDs: AMLSG18-12
Record Dates: First submitted 2012-10-09; First posted 2013-01-17 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia (AML); Histamine Dihydrochloride; Interleukin-2
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a non-interventional multi-center study (NIS) in adult patients with AML in first complete remission with measurable minimal residual disease (MRD). Patients are eligible when gene status was already determined for previous induction and consolidation therapy of AML and showed carrier of NPM1, CBFβ-MYH11, or MLL-AF9 mutation. The study objective is to observe the impact of pre-emptive therapy with histamine dihydrochloride (HDC) and interleukin-2 (IL-2) with regard to assess leukemia-free survival/time to relapse and to monitor MRD level trend over time. HDC and IL-2 are approved drugs for AML patients in first complete remission. Therapy is administered for 10 treatment cycles as outlined in the Summary of Product Characteristics.

ELIGIBILITY:
Patient eligibility criteria in accordance to the summary of Product Characteristics:

* Patients with confirmed diagnosis of acute myeloid leukemia according to the World Health Organization (WHO) classification (including de novo AML, t-AML and s-AML) in first complete remission (defined as less than 5% blasts in a normocellular bone marrow assessed prior to the treatment start)
* AMLSG BiO participation incl. favourable opinion
* Presence of NPM1 mutation, CBFB-MYH11 or MLL-AF9 fusion genes as assessed in one of the central AMLSG reference laboratories.
* Measurable MRD values (non-negative values after consolidation therapy or increase in values over the threshold during follow-up in complete remission)
* The patient must be informed of the observation and written informed consent regarding data privacy obtained.
* Consent for registration, storage and processing of the individual disease-characteristics and course as well as information of the family physician and all other treating physicians about observation participation
* No continuing systemic treatment with clonidine, steroids, and/or H2 receptor blocking agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute myeloid leukaemia (AML) in first remission following completion of consolidation therapy and concomitantly treated with interleukin-2 (IL-2) which will receive treatment with CEPLENE® for the first time. Patients are eligible when gene status was already determined for previous induction and consolidation therapy of AML and showed carrier of NPM1, CBFβ-MYH11, or MLL-AF9 mutation.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-10; Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
leukemia-free survival / cumulative incidence of relapse | two years

SECONDARY OUTCOMES:
Toxicity induced by the preemptive treatment with Ceplene and IL-2 | 18 months
  Duration of neutropenia and leukopenia after each treatment cycle, incidence of infections, duration of hospitalization
Overall survival | two years

OTHER OUTCOMES:
Assessment of quality of life | two years

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Greiner, MD, Principal Investigator — University Hospital of Ulm
Locations (22):
- Germany (22):
  - Vivantes Hospital Neukölln, Berlin
  - Charite, University Medical School of Berlin, Berlin
  - Darmstadt Clinic, Darmstadt
  - University Hospital of Düsseldorf, Düsseldorf
  - Malteser Krankenhaus St. Franziskus Hospital, Flensburg
  - University of Freiburg, Freiburg im Breisgau
  - Wilhelm-Anton-Hospital gGmbH Goch, Goch
  - Klinikum Region Hannover GmbH, Krankenhaus Siloah, Hanover
  - Hannover Medical School, Hanover
  - Saarland University Medical Center, Homburg/Saar
  - Städtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - University Medical Center Schleswig Holstein, Kiel
  - Caritas-Krankenhaus Lebach, Lebach
  - Hospital of Lüdenscheid, Lüdenscheid
  - University Clinic Magdeburg, Magdeburg
  - Hospital of Schwäbisch Gmünd, Mutlangen
  - University Hospital rechts der Isar, München
  - Hospital of Passau, Passau
  - Hospital of Traunstein, Traunstein
  - Klinikum Mutterhaus der Borromäerinnen, Trier
  - University Hospital of Ulm, Ulm
  - Helios Klinikum Wuppertal, Wuppertal